CLINICAL TRIAL: NCT04693455
Title: A Phase 1, Double Blind, Randomized, Placebo Controlled, Single Dose, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZD03 Capsule in Healthy Volunteers in The United States
Brief Title: ZD03 Capsule Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanxi Zhendong Leading Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanxi Zhendong Pharmacy Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ZDXD-ZD03-US-19-4
Record Dates: First submitted 2020-12-01; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Experimental: Cohort 1, Dose 1 of ZD03 or Placebo (Experimental): Dose 1 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo
- Experimental: Cohort 2, Dose 2 of ZD03 or Placebo (Experimental): Dose 2 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo
- Experimental: Cohort 3, Dose 3 of ZD03 or Placebo (Experimental): Dose 3 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo
- Experimental: Cohort 4, Dose 4 of ZD03 or Placebo (Experimental): Dose 4 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo
- Experimental: Cohort 5, Dose 5 of ZD03 or Placebo (Experimental): Dose 5 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo
- Experimental: Cohort 6, Dose 6 of ZD03 or Placebo (Experimental): Dose 6 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo
- Experimental: Cohort 7, Dose 7 of ZD03 or Placebo (Experimental): Dose 7 of ZD03 or matching Placebo capsules by mouth
  Interventions: Drug: ZD03; Other: Placebo

INTERVENTIONS:
Drug: ZD03 — ZD03 capsule
Other: Placebo — placebo capsule

SUMMARY:
This is a Phase 1, Double Blind, Randomized, Placebo Controlled, Single Dose, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZD03 Capsule in Healthy Volunteers in The United States

DETAILED DESCRIPTION:
ZD03 is a novel small molecular drug. It is a synthetic chemical drug candidate for treatment of multiple sclerosis (MS) and is proposed to be administered orally as capsules.

This is a double-blind, randomized, placebo-controlled, single ascending dose study. Approximately 56 HVs will enter into the phase 1 study. The study is designed to evaluate the safety,tolerability and PK of ZD03 capsule at different dose cohorts when administered orally.

Subjects who meet the enrollment criteria will be enrolled in one of the seven dose levels designated for the study, including the doses of 20, 40, 80, 120, 180, 240 and 300 mg (doses escalated by 100%, 100%, 50%, 50%, 33% and 25%, respectively). Each cohort will consist of 8 subjects randomized at 3:1 to receive a single oral dose of ZD03 (n=6) or placebo (n=2) in a double-blind manner in a fasted state

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18 to 55 years, inclusive.
2. An attempt will be made to recruit at least 50% non-Hispanic Caucasians in each cohort,Healthy (no clinically significant health concerns), as determined by medical history, physical examination, 12-lead ECG, and vital signs at screening.
3. Subjects must have a Body Mass Index (BMI) between 18.0 and 30.0 kg/m2 at screening (inclusive) and weighed a minimum of 50 kg (110 lbs).
4. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal ligation, Essure procedure, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or postmenopausal for ≥ 12 months. The site will attempt to retrieve medical records to document sterility; however, the absence of records will not exclude screening the subject. If medical records cannot be obtained, a negative pregnancy test at screening will be accepted. Postmenopausal status will be confirmed through testing of FSH (follicle stimulating hormone) levels by PI discretion at screening for amenorrhoeic female subjects.

   Males must be surgically sterile (> 30 days since vasectomy with no viable sperm), abstinent or if engaged in sexual relations with a female partner of child-bearing potential, the subject must be using a condom with spermicide from Screening and for a period of 30 days after the last dose of Study Drug.

   Acceptable methods of contraception for males are condoms with spermicide.
5. Subjects must have a complete blood count (CBC) and platelet count within the normal range or considered not clinically significant by the PI.
6. Subjects must have normal blood chemistry or results considered not clinically significant by the investigator including electrolytes (Na+, K+, Ca++, and Cl-), alkaline phosphatase, total protein, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, uric acid, creatinine, blood urea nitrogen (BUN), and glucose.
7. Subjects must have a normal urinalysis or results considered not clinically significant by the investigator including a normal protein/creatinine ratio per local lab reference ranges (< 200 mg/g) and a urine creatinine result that does not exceed 300 mg/dL.
8. Subjects must have estimated glomerular filtration rate (eGFR) ≥ 90 mL/min(Based on MDRD).
9. Subjects must have a normal ECG or results considered not clinically significant by the PI.
10. Subjects must be able to comply with the study and follow-up procedures.
11. Subjects are able to understand the study procedures and risks involved and must provide signed informed consent to participate in the study

Exclusion Criteria:

1. Subjects with any history or clinical manifestations of significant metabolic, hematological, pulmonary, including latent tuberculosis, cardiovascular, gastrointestinal including cholecystectomy, neurologic, hepatic, renal, urological, or psychiatric disorders.
2. Subjects who have any history or suspicion of kidney stones.
3. Subjects who are positive for human immunodeficiency virus (HIV), Hepatitis B surface antigen, Hepatitis C virus, and/or treponema pallidum.
4. Subjects who have used prescription drugs, over-the-counter drugs, or herbal remedies within 14 days before Day 1 of study medication dosing. Females who have received hormone replacement therapy (HRT) within 28 days prior to dosing.
5. Subjects who have undergone major surgery within 3 months prior to Day 1.
6. Women who are pregnant or breastfeeding.
7. Subjects who received any investigational test article within 5 half-lives or 30 days, whichever is longer, prior to Day 1 study medication dosing.
8. Subjects who consumed Seville oranges or grapefruit containing foods or beverages within 7 days before Day 1 and during the entire study duration.
9. Subjects who had been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may have impacted subject safety or the validity of the study results.
10. Subjects who had a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine.
11. Subjects with any condition that, in the judgment of the investigator, would place him/her at undue risk, or potentially compromise the results or interpretation of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | Up to 14 days
  Safety and tolerability will be assessed by monitoring adverse events (AEs), several adverse events (SAEs)
Number of participants with clinically significant Vital sign abnormalities will be assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 | Screening, Day -1 to Day 1, Day 2 and Day 7
  Assessed as number of participants with clinically significant changes from Baseline, compared across arms. Vital signs including sitting blood pressure, pulse rate, respiration rate and oral temperature.
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities will be assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 | Screening, Day -1 to Day 1, Day 2 and Day 7
  Assessed as number of participants with clinically significant changes from Baseline, compared across arms. Resting 12-lead ECGs will use a standard 12-lead ECG machine that automatically calculates HR and measures RR, PR, QRS, QT and QTc intervals.
Number of participants with clinically significant physical examination abnormalities will be assessed by discretion of the investigator | Screening, Day -1 to Day 1, Day 2 and Day 7
  Assessed as number of participants with clinically significant changes from Baseline, compared across arms. Physical examination including the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities.
Number of participants with clinically significant haematology assessment abnormalities will be assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 | Screening, Day -1 to Day 1, Day 2 and Day 7
  Assessed as number of participants with clinically significant changes from Baseline, compared across arms. Haematology including Basophils (abs), Eosinophils (abs), Hemoglobin, Monocytes (abs), Neutrophils (abs), Platelets, RBC and WBC, etc.
Number of participants with clinically significant serum chemistry assessment abnormalities will be assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 | Screening, Day -1 to Day 1, Day 2 and Day 7
  Assessed as number of participants with clinically significant changes from Baseline, compared across arms. Serum chemistry including Magnesium, Albumin, Phosphorus, Potassium, Sodium, Total Bilirubin, Total Protein, and Triglyceride, etc.
Number of participants with clinically significant urinalysis assessment abnormalities will be assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 | Screening, Day -1 to Day 1, Day 2 and Day 7
  Assessed as number of participants with clinically significant changes from Baseline, compared across arms. Urinalysis including Bilirubin, Clarity, Color, Glucose, Ketone, Leukocyte, esterase, Protein, Specific, gravity, and Urobilinogen, etc.

SECONDARY OUTCOMES:
PK parameters-AUC0-t | Up to 24 hours
  area under the concentration-time curve from time 0 to the time of last quantifiable concentration (tlast), calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations
PK parameters-AUC0-∞ | Up to 24 hours
  area under the concentration-time curve from time 0 extrapolated to infinity
PK parameters-Cmax | Up to 24 hours
  maximum observed plasma concentration
PK parameters-tmax | Up to 24 hours
  time of maximum observed plasma concentration
PK parameters-t1/2 | Up to 24 hours
  apparent plasma terminal elimination half-life
PK parameters-CL/F | Up to 24 hours
  apparent total plasma clearance
PK parameters-Vz/F | Up to 24 hours
  apparent volume of distribution during the terminal elimination phase

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials,Early Phase Services, LLC, San Antonio, Texas, United States